CLINICAL TRIAL: NCT00454896
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Assess the Efficacy and Safety of Daily Oral Administration of 5mg and 10mg VESIcare® for the Treatment of Urgency Associated With Overactive Bladder
Brief Title: A Multicenter VESIcare® Efficacy and Safety Study for the Treatment of Urgency Associated With Overactive Bladder (OAB)
Acronym: VENUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 905-UC-005
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urinary Bladder, Overactive; Urgency; VESIcare®; Solifenacin succinate
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: VESIcare®
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: VESIcare® — Oral
  Other Names: solifenacin succinate; YM905
  Arms: 1
Drug: placebo — Oral
  Arms: 2

SUMMARY:
The purpose is to evaluate the efficacy of 5 and 10mg VESIcare® (solifenacin succinate) in patients with urgency who have overactive bladder syndrome.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 urinary urgency episode/24h (on average) documented in a 3-day patient diary in the screening phase with or without urge incontinence, and usually with frequency and nocturia, described as OAB
* Patients may be included if they were never exposed to anticholinergic agents specified for the treatment of OAB. Patients may also be included if they have previously been treated with FDA-approved anticholinergic agents for the treatment of OAB such as oxybutynin chloride and are no longer receiving such treatment for a minimum of 14 days immediately preceding entry into the study. These previously treated patients must present at the investigative site on no anticholinergic agents and with the desire to receive treatment for OAB. Previous non-drug treatment of OAB is allowed if it has been established at least 4 weeks prior to study entry and is continued throughout the study.
* Patients having urgency with or without urge incontinence accompanied by frequency of ≥8 episodes per 24 hours, and/or nocturia, for a period of ≥3 months prior to screening.

Exclusion Criteria:

* Previous treatment with darifenacin
* Duration of urgency with or without urge incontinence, usually accompanied with frequency and nocturia for <3 months
* Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor as determined by the Investigator
* Evidence of a urinary tract infection; chronic inflammation such as interstitial cystitis and bladder stones
* Clinically significant outflow obstruction (benign prostatic hyperplasia) as determined by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2004-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of 5 and 10mg solifenacin succinate in patients with urgency who have OAB syndrome | Weeks 1, 4, 8 and 12

SECONDARY OUTCOMES:
Improvement of urgency | Weeks 1, 4, 8 and 12
Improvement of frequency, incontinence and nocturia | Weeks 1, 4, 8 and 12
Number of patients satisfied with treatment | Weeks 1, 4, 8 and 12
Assessment of the efficacy | End of study
Evaluation of the safety and tolerability | Baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (63):
- United States (63):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Atherton, California
  - Carmichael, California
  - Escondido, California
  - Fresno, California
  - Los Angeles, California
  - Mission Hills, California
  - Mission Viejo, California
  - Salinas, California
  - Valley Village, California
  - Aurora, Colorado
  - Denver, Colorado
  - New London, Connecticut
  - Norwalk, Connecticut
  - Trumbull, Connecticut
  - Waterbury, Connecticut
  - Washington D.C., District of Columbia
  - Boyton Beach, Florida
  - Clearwater, Florida
  - Gainesville, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Tallahassee, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Blue Ridge, Georgia
  - Marietta, Georgia
  - Boise, Idaho
  - Centralia, Illinois
  - Slidell, Louisiana
  - Bloomfield Hills, Michigan
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Lawrenceville, New Jersey
  - South Bound Brook, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - East Syracuse, New York
  - Hewlett, New York
  - Lewiston, New York
  - New York, New York
  - Concord, North Carolina
  - Hickory, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Eugene, Oregon
  - Endwell, Pennsylvania
  - Media, Pennsylvania
  - Monroeville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Uniontown, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Athens, Texas
  - Ogden, Utah
  - West Point, Utah
  - Richmond, Virginia
  - Spokane, Washington
  - Vancouver, Washington
  - Morgantown, West Virginia

REFERENCES:
- [Background] Karram MM, Toglia MR, Serels SR, Andoh M, Fakhoury A, Forero-Schwanhaeuser S. Treatment with solifenacin increases warning time and improves symptoms of overactive bladder: results from VENUS, a randomized, double-blind, placebo-controlled trial. Urology. 2009 Jan;73(1):14-8. doi: 10.1016/j.urology.2008.08.485. Epub 2008 Nov 8. PMID 18995887
- [Background] Toglia MR, Serels SR, Laramee C, Karram MM, Nandy IM, Andoh M, Seifeldin R, Forero-Schwanhaeuser S. Solifenacin for overactive bladder: patient-reported outcomes from a large placebo-controlled trial. Postgrad Med. 2009 Sep;121(5):151-8. doi: 10.3810/pgm.2009.09.2062. PMID 19820284
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Serels SR, Toglia MR, Forero-Schwanhaeuser S, He W. Impact of solifenacin on diary-recorded and patient-reported urgency in patients with severe overactive bladder (OAB) symptoms. Curr Med Res Opin. 2010 Oct;26(10):2277-85. doi: 10.1185/03007995.2010.509582. PMID 20707767